CLINICAL TRIAL: NCT05903521
Title: Long-term Impact of Surgically Induced Rapid Weight Loss on Telomere Length and Its Potential Implications in the Genesis and Prevention of Neoplastic Disease Processes in Subjects With Severe Obesity
Brief Title: BAriatric Surgery Induced Chromosomal Change
Acronym: BASICC
Status: Terminated | Type: Observational
Why Stopped: Issue with telomere measurement
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Emanuele LoMenzo, Prof., The Cleveland Clinic
Other Study IDs: 23-488
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Obesity, Morbid
Keywords: Telomere length; Metabolic and bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: BMI ≥ 35 kg/m2 without previous bariatric surgery
- Treatment group: Having had Sleeve Gastrectomy or Roux-en-Y Gastric Bypass more than 12 months ago and without a weight regain of ≥ 15% of nadir weight

SUMMARY:
The purpose of this study is to better understand the impact of weight-loss surgery on telomere length. Telomeres are a key marker of biological aging of cells. Telomere shortening is a natural process of aging. Several pathologies and lifestyles are associated with premature telomere shortening, such as obesity, diabetes mellitus or sedentary lifestyle. New evidence supports that telomere shortening can be partially reversed by lifestyle changes such as healthy diet, reduced stress, or increased physical activity.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of metabolic and bariatric surgery on telomere length as well as the role of type 2 diabetes resolution and oxidative stress improvement on telomere lengthening.

The investigators hypothesize that metabolic and bariatric surgery is associated with the lengthening of telomeres as a possible underlying mechanism of cancer risk reduction.

It is a prospective, single-center study including patients with obesity class II or more (Body Mass Index ≥ 35kg/m2) and patients having had metabolic and bariatric surgery more than 12 months ago.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m2 without previous bariatric surgery (control group) OR
* Having had Sleeve Gastrectomy or Roux-en-Y Gastric Bypass more than 12 months ago and without a weight regain of ≥ 15% of nadir weight (treatment group)

Exclusion Criteria:

* under 18 years of age
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be divided in two groups; the control group (with obesity) and the treatment group (after Sleeve Gastrectomy or Roux-en-Y Gastric Bypass).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Telomere length | 1 day
  Difference in terms of telomere length between patients with obesity class II or more (Body Mass Index [BMI] ≥ 35kg/m2) and patients after metabolic and bariatric surgery.

SECONDARY OUTCOMES:
Metabolic disease remission (hypertension and type 2 diabetes remission versus no remission) | 1 day
  Evaluate if remission of metabolic disease (no remission versus remission) has an impact of metabolic disease remission on telomere length after bariatric and metabolic surgery
Excessive weight loss (Weight loss [kg] / excess body weight [kg]) x 100 = Percent of excess body weight loss) | 1 day
  Evaluate if the amount of excessive weight loss has an impact on telomere length after bariatric and metabolic
Lifestyle (Simple Lifestyle Indicator Questionnaire) | 1 day
  Evaluate if lifestyle (Simple Lifestyle Indicator Questionnaire) has an impact of lifestyle on telomere length after bariatric and metabolic
Oxidative stress (Interleukin-1β, Interleukin-6, TNF-α) | 1 day
  Evaluate if oxidative stress level (Interleukin-1β, Interleukin-6, TNF-α) has an impact on telomere length after bariatric and metabolic

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No